CLINICAL TRIAL: NCT04180163
Title: A Phase 3 Multi-center, Open-label Study to Evaluate the Efficacy and Safety of Lanadelumab (SHP643) in Japanese Subjects With Hereditary Angioedema
Brief Title: Efficacy and Safety of Lanadelumab (SHP643) in Japanese Participants With Hereditary Angioedema (HAE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP643-302; 195014 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Results first posted 2022-09-19 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — lanadelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lanadelumab 300 mg q2w or q4w (Experimental): Lanadelumab 300 mg solution, subcutaneously (SC), once every 2 weeks (q2w) for 26 weeks in Treatment Period A. This was followed by Treatment Period B (additional 26 weeks, total of 52 weeks including Treatment Period A) during which participants remained on Treatment Period A regimen or received 300 mg lanadelumab solution once every 4 weeks (q4w) for 26 weeks if well-controlled (attack-free) for 26 consecutive weeks with lanadelumab treatment. The dose frequency change was based on the Investigator's discretion and approval by the Sponsor's Medical Monitor.
  Interventions: Drug: Lanadelumab

INTERVENTIONS:
Drug: Lanadelumab — Lanadelumab solution, SC
  Other Names: DX-2930; TAK-743; SHP643

SUMMARY:
The purpose of this phase 3, open-label, multi-center study is to evaluate the safety and efficacy of lanadelumab in Japanese participants with HAE Type I or II.

DETAILED DESCRIPTION:
This study will consist of 52-week treatment period and a 4-week follow-up period. 52-week treatment period comprises of a 26-week treatment period A (Day 0 to Day 182) and a 26-week treatment period B (Day 183 to Day 364). Participants who complete treatment period A will immediately continue into treatment period B. After completion of treatment period B participants may roll over into an expanded access study TAK-743-5007 (NCT04687137). Participants who elect to rollover to Study TAK-743-5007 will complete their end of study (EOS) assessments on Day 378. All other participants will complete their EOS assessments on Day 392.

ELIGIBILITY:
Inclusion Criteria:

* Be of Japanese descent, defined as born in Japan and having Japanese parents and Japanese maternal and paternal grandparents.
* The participant is male or female and >= 12 years of age at the time of informed consent.
* Documented diagnosis of HAE (Type I or II) based upon all of the following:

  1. Documented clinical history consistent with HAE (subcutaneous or mucosal, nonpruritic swelling episodes without accompanying urticaria).
  2. Diagnostic testing results obtained during screening that confirm HAE Type I or II: C1 inhibitor (C1-INH) functional level <40% of the normal level. Participants with functional C1-INH level 40-50% of the normal level may be enrolled if they also have a C4 level below the normal range. With prior sponsor approval, participants may be retested during the run-in period if results are in congruent with clinical history or believed by the investigator to be confounded by recent C1 inhibitor use.
  3. At least one of the following: age at reported onset of first angioedema symptoms <=30 years, a family history consistent with HAE Type I or II, or C1q within normal range.
* Attack rate: Participants must experience at least 1 investigator-confirmed HAE attack per 4 weeks during the run-in period to enter the lanadelumab treatment period.
* The participant (or the participants parent/legal authorized representative, if applicable) has provided written informed consent approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC).
* If the participant is an adult, be informed of the nature of the study and provide written informed consent before any study-specific procedures are performed or if the participant is a minor (ie, below the age of majority), have a parent/legally authorized representative who is informed of the nature of the study provide written informed consent (ie, permission) for the minor to participate in the study before any study-specific procedures are performed. Assent will be obtained from minor participants.
* Males, or non pregnant, non lactating females who are fertile and sexually active and who agree to be abstinent or agree to comply with the applicable contraceptive requirements of this protocol for the duration of the study, or females of non child bearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or postmenopausal for at least 12 months.
* Agree to adhere to the protocol-defined schedule of assessments and procedures.

Exclusion Criteria:

* Concomitant diagnosis of another form of chronic, recurrent angioedema, such as acquired angioedema (AAE), HAE with normal C1-INH (also known as HAE Type 3), idiopathic angioedema, or recurrent angioedema associated with urticaria.
* Participation in a prior lanadelumab study.
* Dosing with investigational drug or exposure to an investigational device within 4 weeks prior to entering to screening.
* Exposure to angiotensin-converting enzyme (ACE) inhibitors or any estrogen-containing medications with systematic absorption (such as oral contraceptives or hormonal replacement therapy) within 4 weeks prior to screening.
* Exposure to androgens (eg, danazol, methyltestosterone, testosterone) within 2 weeks prior to entering the run-in period.
* Use of long-term prophylactic therapy for HAE (C1-INH, attenuated androgens, or anti-fibrinolytics) within 2 weeks prior to entering the run in period.
* Use of short-term prophylaxis for HAE 7 days prior to entering the run-in period. Short-term prophylaxis is defined as C1-INH, attenuated androgens, or anti-fibrinolytics used to avoid angioedema complications from medically indicated procedures.
* Any of the following liver function abnormalities: alanine aminotransferase (ALT) >3x upper limit of normal, or aspartate aminotransferase (AST) >3x upper limit of normal or bilirubin >2x upper limit of normal (unless the bilirubin is a result of Gilbert's syndrome).
* Pregnancy or breast feeding.
* Participant has any condition that in the opinion of the investigator or sponsor, may compromise their safety or compliance, preclude successful conduct of the study, or interfere with interpretation of the results (eg, history of substance abuse, or dependence, significant preexisting illnesses or major comorbidity the investigator considers may confound the interpretation of the study results).
* Participant has a known hypersensitivity to the IP or its components.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- Japan (12):
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Asahi General Hospital, Asahi-shi, Chiba
  - Ogaki Municipal Hospital, Ogaki-shi, Gifu
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Tomakomai City Hospital, Tomakomai-shi, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Tokai University Hospital, Isehara-shi, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Kyoto University Hospital, Kyoto, Kyoto
  - Osaka University Hospital, Suita-shi, Osaka
  - Saiyu Soka Hospital, Soka-shi, Saitama
  - Shimane University Hospital, Izumo-shi, Shimane

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fdc4db2bf003ab472fb

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 participants took part in the study at 10 investigative sites in Japan from 12 December 2019 to 26 August 2021.
Pre-assignment Details: Enrolled participants were observed in 4-week Baseline Run-in Period that could be extended up to 8 weeks. Participants who experienced ≥1.0 angioedema attacks per 4 weeks during the Run-in Period and who remained eligible per inclusion criteria entered 52-week lanadelumab Treatment Period (Treatment Period A + Treatment Period B), followed by up to 4-week Safety Follow-up Period. Participants received lanadelumab only during the Treatment Periods.
Period: Run-in Period (4 or up to 8 Weeks)
Arm/Group | Lanadelumab 300 mg q2w or q4w
Started | 12
Completed | 12
Not Completed | 0
Period: Treatment Period A (Weeks 1 to 26)
Arm/Group | Lanadelumab 300 mg q2w or q4w
Started | 12
Completed (Completion of Treatment Period A was defined as completion of any of the Day 182 visit assessments.) | 12
Not Completed | 0
Period: Treatment Period B (Weeks 27 to 52)
Arm/Group | Lanadelumab 300 mg q2w or q4w
Started | 12
Completed (Completion of Treatment Period B was defined as completion of any of the Day 364 visit assessments.) | 12
Not Completed | 0
Period: Safety Follow-up Period (Weeks 53 to 56)
Arm/Group | Lanadelumab 300 mg q2w or q4w
Started (Participants who rolled over to TAK-743-5007 (NCT04687137) had a 2-week follow-up while others had 4 weeks of follow-up.) | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of investigational medicinal product (IMP).
Groups:
- Lanadelumab 300 mg q2w or q4w: Lanadelumab 300 mg solution, SC, q2w for 26 weeks in Treatment Period A. This was followed by Treatment Period B (additional 26 weeks, total of 52 weeks including Treatment Period A) during which participants remained on Treatment Period A regimen or received 300 mg lanadelumab solution q4w for 26 weeks if well-controlled (attack-free) for 26 consecutive weeks with lanadelumab treatment. The dose frequency change was based on the Investigator's discretion and approval by the Sponsor's Medical Monitor.
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 12
Weight [Mean (Standard Deviation); unit: kg] | 61.24 (10.346)
Height [Mean (Standard Deviation); unit: cm] | 161.08 (9.379)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI= weight(kg) / height(meter)^2
  kg/m^2 | 23.80 (5.065)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Attack-Free Status for the Efficacy Evaluation Period of Day 0 Through Day 182
Description: A participant was considered as attack free during an efficacy evaluation period if the participant had no investigator-confirmed hereditary angioedema (HAE) attacks during that efficacy evaluation period. A HAE attack was defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). Number of participants achieving attack-free status for the efficacy evaluation period of Day 0 through Day 182 were assessed.
Time Frame: Day 0 through Day 182
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
Participants | 5

2. Secondary Outcome: Number of Investigator-Confirmed Hereditary Angioedema (HAE) Attacks During Each of the Efficacy Evaluation Periods
Description: Efficacy evaluation period consisted of four periods: Day 0 (after study drug administration) through Day 182 (the end of Treatment Period A), Day 0 (after study drug administration) through Day 364 (the end of Treatment Period B), presumed steady-state period from Day 70 through Day 182, presumed steady-state period from Day 70 through Day 364. Number of investigator-confirmed HAE attacks during each of the efficacy evaluation periods were assessed.
Time Frame: Day 0 through Day 182, Day 0 through Day 364, Day 70 through Day 182, Day 70 through Day 364
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Number; unit: HAE attacks
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
HAE attacks
  Day 0 Through Day 182 | 92
  Day 0 Through Day 364 | 189
  Day 70 Through Day 182 | 55
  Day 70 Through Day 364 | 152

3. Secondary Outcome: Number of Investigator-Confirmed Hereditary Angioedema (HAE) Attacks Requiring Acute Treatment During Each of the Efficacy Evaluation Periods
Description: Efficacy evaluation period consisted of four periods: Day 0 (after study drug administration) through Day 182 (the end of Treatment Period A), Day 0 (after study drug administration) through Day 364 (the end of Treatment Period B), presumed steady-state period from Day 70 through Day 182, presumed steady-state period from Day 70 through Day 364. Number of investigator-confirmed HAE attacks requiring acute treatment during each of the efficacy evaluation periods were assessed.
Time Frame: Day 0 through Day 182, Day 0 through Day 364, Day 70 through Day 182, Day 70 through Day 364
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Number; unit: HAE attacks
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
HAE attacks
  Day 0 Through Day 182 | 79
  Day 0 Through Day 364 | 168
  Day 70 Through Day 182 | 46
  Day 70 Through Day 364 | 135

4. Secondary Outcome: Number of Moderate or Severe Investigator-Confirmed Hereditary Angioedema (HAE) Attacks During Each of the Efficacy Evaluation Periods
Description: Severe attack was defined as Grade 3 (some assistance usually required, medical intervention/therapy required, hospitalizations possible), moderate attack was defined as Grade 2 (some assistance may be needed, no or minimal medical intervention/therapy required). Number of investigator-confirmed moderate or severe HAE attacks during the each of efficacy evaluation periods was assessed. Efficacy evaluation period consisted of four periods: Day 0 (after study drug administration) through Day 182 (the end of Treatment Period A), Day 0 (after study drug administration) through Day 364 (the end of Treatment Period B), presumed steady-state period from Day 70 through Day 182, presumed steady-state period from Day 70 through Day 364.
Time Frame: Day 0 through Day 182, Day 0 through Day 364, Day 70 through Day 182, Day 70 through Day 364
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Number; unit: HAE attacks
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
HAE attacks
  Day 0 Through Day 182 | 72
  Day 0 Through Day 364 | 153
  Day 70 Through Day 182 | 41
  Day 70 Through Day 364 | 122

5. Secondary Outcome: Number of Participants With Maximum Hereditary Angioedema (HAE) Attack Severity During Each of the Efficacy Evaluation Periods
Description: Efficacy evaluation period consisted of four periods: Day 0 (after study drug administration) through Day 182 (the end of Treatment Period A), Day 0 (after study drug administration) through Day 364 (the end of Treatment Period B), presumed steady-state period from Day 70 through Day 182, presumed steady-state period from Day 70 through Day 364. Number of participants with maximum HAE attack severity during each of the efficacy evaluation periods was assessed. HAE attack severity was calculated per participant based on the severity categories as follows: No attack, Mild, Moderate, and Severe.
Time Frame: Day 0 through Day 182, Day 0 through Day 364, Day 70 through Day 182, Day 70 through Day 364
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
Participants
  Day 0 Through Day 182: No Attack | 5
  Day 0 Through Day 182: Mild | 2
  Day 0 Through Day 182: Moderate | 4
  Day 0 Through Day 182: Severe | 1
  Day 0 Through Day 364: No Attack | 2
  Day 0 Through Day 364: Mild | 1
  Day 0 Through Day 364: Moderate | 8
  Day 0 Through Day 364: Severe | 1
  Day 70 Through Day 182: No Attack | 5
  Day 70 Through Day 182: Mild | 4
  Day 70 Through Day 182: Moderate | 2
  Day 70 Through Day 182: Severe | 1
  Day 70 Through Day 364: No Attack | 2
  Day 70 Through Day 364: Mild | 2
  Day 70 Through Day 364: Moderate | 7
  Day 70 Through Day 364: Severe | 1

6. Secondary Outcome: Number of High-Morbidity Investigator-Confirmed Hereditary Angioedema (HAE) Attacks During Each of the Efficacy Evaluation Periods
Description: A high morbidity HAE attack was defined as any attack that has at least 1 of the following characteristics: severe, results in hospitalization (except hospitalization for observation <24 hours), hemodynamically significant (systolic blood pressure <90, requires intravenous (IV) hydration, or associated with syncope or near syncope) or laryngeal. Number of high-morbidity investigator-confirmed HAE attacks during each of the 4 efficacy evaluation periods (Treatment Period A, Overall Treatment Period, Presumed Steady-state Period for Treatment Period A and Overall Presumed Steady-state Period) were assessed.
Time Frame: Day 0 through Day 182, Day 0 through Day 364, Day 70 through Day 182, Day 70 through Day 364
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Number; unit: HAE attacks
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
HAE attacks
  Day 0 Through Day 182 | 5
  Day 0 Through Day 364 | 11
  Day 70 Through Day 182 | 4
  Day 70 Through Day 364 | 10

7. Secondary Outcome: Time to First Hereditary Angioedema (HAE) Attack After Day 0 for the Efficacy Evaluation Period
Description: The time to the first HAE attack (days) after Day 0 for the efficacy evaluation period of Day 0 through Day 182 was calculated from the date and time of the first dose of lanadelumab for the efficacy evaluation period (Day 0 through Day 182) to the date and time of the first in HAE attack after the first open-label dose for the efficacy evaluation period of Day 0 through Day 182. Kaplan-Meier Method was used for analysis and the Kaplan Meier estimate expressed as time (in days) to first HAE attack After Day 0 for Treatment Period A (Day 0 through Day 182) is presented.
Time Frame: Day 0 through Day 182
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
days | 97.2 [4.2 to NA] — The upper limit of 95% confidence interval (CI) was not evaluable due to low number of participants with events.

8. Secondary Outcome: Time to First Hereditary Angioedema (HAE) Attack After Day 0 for the Efficacy Evaluation Period
Description: The time to the first HAE attack (days) after Day 0 for the efficacy evaluation period of Day 70 through Day 182 was calculated from the date and time of the first dose of lanadelumab for the efficacy evaluation period (Day 70 through Day 182) to the date and time of the first in HAE attack after the first open-label dose for the efficacy evaluation period of Day 70 through Day 182. Kaplan-Meier Method was used for analysis and the Kaplan Meier estimate expressed as time (in days) to first HAE attack After Day 0 for presumed steady-state period for Treatment Period A (Day 70 through Day 182) is presented.
Time Frame: Day 70 through Day 182
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
days | 91.0 [4.6 to NA] — The upper limit of 95% CI was not evaluable due to low number of participants with events.

9. Secondary Outcome: Number of Participants Achieving at Least 50%, 70% and 90% Reduction in the Investigator-Confirmed Normalized Number of Attacks (NNA) Per 4 Weeks Relative to the Run-in Period NNA for Each of Efficacy Evaluation Periods
Description: Run- in Period was 4 weeks and may have been extended up to 8 weeks to determine participants' Baseline attack rate. The normalized number of investigator-confirmed HAE attacks (NNA) during each efficacy evaluation period will be expressed as a monthly (28 days) HAE attack rate. Number of participants achieving at least 50%, 70% and 90% reduction in the investigator-confirmed NNA per 4 weeks relative to the Run-in Period normalized NNA for each of the 4 efficacy evaluation periods (Treatment Period A, Overall Treatment Period, Presumed Steady-state Period for Treatment Period A, and Overall Presumed Steady-state Period) were assessed. For each participant, the percentage reduction was calculated as the run-in period attack rate minus the treatment period attack rate divided by the run-in period attack rate, multiplied by 100. The responder categories were not mutually exclusive, participants may appear in more than one category as applicable based on their percentage reduction.
Time Frame: Day 0 through Day 182, Day 0 through Day 364, Day 70 through Day 182, Day 70 through Day 364
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
Participants
  Day 0 Through Day 182: ≥50% Reduction | 10
  Day 0 Through Day 182: ≥70% Reduction | 8
  Day 0 Through Day 182: ≥90% Reduction | 6
  Day 0 Through Day 364: ≥50% Reduction | 10
  Day 0 Through Day 364: ≥70% Reduction | 8
  Day 0 Through Day 364: ≥90% Reduction | 6
  Day 70 Through Day 182: ≥50% Reduction | 11
  Day 70 Through Day 182: ≥70% Reduction | 10
  Day 70 Through Day 182: ≥90% Reduction | 6
  Day 70 Through Day 364: ≥50% Reduction | 10
  Day 70 Through Day 364: ≥70% Reduction | 8
  Day 70 Through Day 364: ≥90% Reduction | 7

10. Secondary Outcome: Number of Participants Achieving Normalized Number of Attacks (NNA) <1.0 Per 4 Weeks, <0.75 Per 4 Weeks, <0.50 Per 4 Weeks and <0.25 Per 4 Weeks for Each of the Efficacy Evaluation Periods
Description: The NNA (investigator-confirmed) during each efficacy evaluation period was expressed as a monthly (28 days) HAE attack rate. Number of participants achieving NNA <1.0 per 4 weeks, <0.75 per 4 weeks, <0.50 per 4 weeks, and <0.25 per 4 weeks for each of the 4 efficacy evaluation periods (Treatment Period A, Overall Treatment Period, Presumed Steady-state Period for Treatment Period A, and Overall Presumed Steady-state Period) were assessed. The responder categories were not mutually exclusive, participants may appear in more than one category as applicable based on their HAE attack rate.
Time Frame: Day 0 through Day 182, Day 0 through Day 364, Day 70 through Day 182, Day 70 through Day 364
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
Participants
  Day 0 Through Day 182: <1.0 per Month | 9
  Day 0 Through Day 182: <0.75 per Month | 9
  Day 0 Through Day 182: <0.50 per Month | 6
  Day 0 Through Day 182: <0.25 per Month | 6
  Day 0 Through Day 364: <1.0 per Month | 9
  Day 0 Through Day 364: <0.75 per Month | 8
  Day 0 Through Day 364: <0.50 per Month | 7
  Day 0 Through Day 364: <0.25 per Month | 6
  Day 70 Through Day 182: <1.0 per Month | 9
  Day 70 Through Day 182: <0.75 per Month | 9
  Day 70 Through Day 182: <0.50 per Month | 8
  Day 70 Through Day 182: <0.25 per Month | 6
  Day 70 Through Day 364: <1.0 per Month | 9
  Day 70 Through Day 364: <0.75 per Month | 8
  Day 70 Through Day 364: <0.50 per Month | 7
  Day 70 Through Day 364: <0.25 per Month | 6

11. Secondary Outcome: Number of Participants Achieving Attack-Free Status for the Efficacy Evaluation Period Day 0 Through Day 364, Day 70 Through Day 182, and Day 70 Through Day 364
Description: A participant was considered as attack free during an efficacy evaluation period if the participant had no investigator-confirmed HAE attacks during that efficacy evaluation period. A HAE attack was defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). Number of participants achieving attack-free status for the 4 efficacy evaluation periods (Overall Treatment Period, Presumed Steady-state Period for Treatment Period A, and Overall Presumed Steady-state Period) were assessed.
Time Frame: Day 0 through Day 364, Day 70 through Day 182, and Day 70 through Day 364
Population: FAS included all participants who received at least 1 dose of IMP. Overall number analyzed are the number of participants who achieved attack-free status during an efficacy evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 9
Participants
  Day 0 Through Day 364 | 2
  Day 70 Through Day 182 | 5
  Day 70 Through Day 364 | 2

12. Secondary Outcome: Number of Participants Achieving Attack-Free Status for Monthly Increments
Description: A participant was considered as attack free during an efficacy evaluation period if the participant had no investigator-confirmed HAE attacks during that efficacy evaluation period. A HAE attack was defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).
Time Frame: At Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 and 13
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
Participants
  Month 1 | 7
  Month 2 | 8
  Month 3 | 9
  Month 4 | 7
  Month 5 | 9
  Month 6 | 7
  Month 7 | 8
  Month 8 | 6
  Month 9 | 7
  Month 10 | 9
  Month 11 | 8
  Month 12 | 7
  Month 13 | 8

13. Secondary Outcome: Number of Participants Achieving Investigator-Confirmed Hereditary Angioedema (HAE) Attack-Free Intervals
Description: A participant was considered as attack free during a time period if the participant had no investigator-confirmed HAE attacks during that time period. Participants who discontinued during a time period were considered as non-responders for that time period. Number of participants achieving investigator-confirmed HAE attack free intervals from Day 0 through Day 182 were assessed.
Time Frame: Day 0 through Day 182
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
Participants | 5

14. Secondary Outcome: Percentage of Attack Free Days During Each of the Efficacy Evaluation Periods
Description: An attack-free day was defined as a calendar day with no investigator-confirmed HAE attack. HAE attack free days were calculated by counting the number of days in the efficacy evaluation period without an HAE attack and dividing by the number of days the participant contributed to the efficacy evaluation period. Percentage of investigator-confirmed HAE attack free days during each of the efficacy evaluation periods (Treatment Period A, Overall Treatment Period, Presumed Steady-state Period for Treatment Period A, and Overall Presumed Steady-state Period) were assessed.
Time Frame: Day 0 through Day 182, Day 0 through Day 364, Day 70 through Day 182, Day 70 through Day 364
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: percentage of attack-free days
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
percentage of attack-free days
  Day 0 Through Day 182 | 88.53 (27.146)
  Day 0 Through Day 364 | 89.04 (27.015)
  Day 70 Through Day 182 | 90.34 (21.952)
  Day 70 Through Day 364 | 89.85 (25.015)

15. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Including Adverse Events of Special Interest (AESI) and Serious Adverse Events (SAEs)
Description: TEAE=any event emerging at or after initiation of treatment with investigational product (IP) or any existing event that worsens in intensity/frequency on exposure to IP. Serious TEAE=any untoward clinical manifestation of signs, symptoms, outcomes (related to IP or not) at any dose: results in death, was life-threatening, requires inpatient/prolongation of hospitalization, resulted in persistent/significant disability/incapacity, congenital abnormality/birth defect, important medical event. AESI=investigator-reported hypersensitivity reactions, events of disordered coagulation as bleeding/hypercoagulable AESI. Adverse events were classified as HAE attack and non-HAE attack reported AEs and are categorized accordingly. As Pre-specified in the protocol, TEAEs, SAEs and AESIs were collected per Period i.e., Treatment Period A, B and Safety follow-up Period and data is reported accordingly.
Time Frame: From first dose of the study drug up to end of study (EOS) (up to Day 392)
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Period A: Non-HAE: Lanadelumab 300 mg solution, SC, q2w for 26 weeks in Treatment Period A. Non-HAE attack (subset identified in case report form [CRF] as not reported HAE attack) subset participants were included in this arm.
- Treatment Period A: HAE: Lanadelumab 300 mg solution, SC, q2w for 26 weeks in Treatment Period A. HAE attack (subset of AEs identified in CRF as reported HAE attack) subset participants were included in this arm.
- Treatment Period B: Non-HAE: Lanadelumab 300 mg solution, SC, q2w for 26 weeks or lanadelumab 300 mg solution, SC, q4w for 26 weeks in Treatment Period B if well tolerated (attack-free) for 26 consecutive weeks with lanadelumab treatment during Treatment Period A. Non-HAE attack (subset identified in CRF as not reported HAE attack) subset participants were included in this arm.
- Treatment Period B: HAE: Lanadelumab 300 mg solution, SC, q2w for 26 weeks or lanadelumab 300 mg solution, SC, q4w for 26 weeks in Treatment Period B if well tolerated (attack-free) for 26 consecutive weeks with lanadelumab treatment during Treatment Period A. HAE attack (subset of AEs identified in CRF as reported HAE attack) subset participants were included in this arm.
- Safety Follow-up Period: Non-HAE: Participants who completed the lanadelumab 300 mg regimen in Treatment Period B returned on Day 378 (for participants who chose to roll over into study TAK-743-5007 [NCT04687137]) or Day 392 as follow-up visit for final assessment in the Safety Follow-up Period. Non-HAE attack (subset identified in CRF as not reported HAE attack) subset participants were included in this arm.
- Safety Follow-up Period: HAE: Participants who completed the lanadelumab 300 mg regimen in Treatment Period B returned on Day 378 (for participants who chose to roll over into study TAK-743-5007) or Day 392 as follow-up visit for final assessment in the Safety Follow-up Period. HAE attack (subset of AEs identified in CRF as reported HAE attack) subset participants were included in this arm.
Arm/Group | Treatment Period A: Non-HAE | Treatment Period A: HAE | Treatment Period B: Non-HAE | Treatment Period B: HAE | Safety Follow-up Period: Non-HAE | Safety Follow-up Period: HAE
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
Participants
  Any TEAEs | 10 [lower limit 111] | 8 | 9 | 8 | 0 | 3
  AESI | 3 [lower limit 34] | 0 | 0 | 0 | 0 | 0
  Any Serious TEAEs | 1 [lower limit 23] | 1 | 1 | 0 | 0 | 0

16. Secondary Outcome: Plasma Concentrations of Lanadelumab
Time Frame: Predose on Days 0, 56, 98, 140, 182, 266, 350, 364, and at any time on Day 378 or 392
Population: Pharmacokinetic (PK) Set included all participants in the FAS who had at least 1 evaluable post dose PK concentration value. Number analyzed is the number of participants available for analysis at a specific time point.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
nanograms per milliliter (ng/mL)
  Day 0 | 25.584 (50.2034)
  Day 56 | 23630.973 (8665.1099)
  Day 98 | 24142.776 (9575.7596)
  Day 140: number analyzed (Participants) | 11
  Day 140 | 24613.885 (9319.6672)
  Day 182 | 23679.526 (6793.3003)
  Day 266 | 19269.249 (8870.0355)
  Day 350: number analyzed (Participants) | 3
  Day 350 | 13225.533 (2538.8239)
  Day 364: number analyzed (Participants) | 10
  Day 364 | 22329.820 (7527.7165)
  Day 378/392 | 19308.033 (7708.1882)

17. Secondary Outcome: Change From Baseline in Angioedema Quality of Life (AE-QoL) Questionnaire Total Score
Description: The AE-QoL questionnaire is a self-administered validated instrument to assess health related (HR)QoL among participants with recurrent angioedema (including HAE). The AE-QoL consists of 17 disease-specific quality-of-life items, to produce a total AE-QoL score and 4 domain scores (functioning, fatigue/mood, fear/shame, and nutrition) and each of the 17 items had a five-point response scale ranging from 1 (Never) to 5 (Very Often). The questionnaire was scored according to the developers' guidelines to produce 4 domain scores (functioning, fatigue/mood, fear/shame, nutrition) yielding a total score. The raw total score (mean of all item scores) was rescaled using linear transformations into final percentage scores ranging 0 to 100, based on the maximum possible score, where higher the score, greater the QoL impairment.
Time Frame: Days 0, 28, 56, 98, 126, 154, 182, 266, 364, 378 or 392
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
score on a scale
  Day 0 | 46.57 (20.885)
  Day 28 | 26.35 (31.129)
  Day 56 | 28.43 (28.255)
  Day 98 | 26.96 (30.926)
  Day 126 | 32.60 (33.999)
  Day 154 | 21.69 (28.750)
  Day 182 | 26.10 (33.978)
  Day 266 | 26.96 (29.951)
  Day 364 | 26.59 (34.428)
  Day 378/392 | 28.55 (31.934)

18. Secondary Outcome: Plasma Kallikrein (pKal) Activity
Description: pKal activity was measured by biomarker cleaved high molecular weight kininogen (cHMWK) level to assess pharmacodynamics (PD) of lanadelumab.
Time Frame: Predose on Days 0, 56, 98, 140, 182, 266, 350, 364, and at any time on Day 378 or 392
Population: Pharmacodynamic (PD) Set included all participants in the FAS who had at least 1 evaluable post dose PD value. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: percentage of cHMWK
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
percentage of cHMWK
  Day 0 | 63.04 (22.096)
  Day 56 | 30.88 (17.090)
  Day 98 | 32.40 (18.829)
  Day 140: number analyzed (Participants) | 11
  Day 140 | 35.67 (13.787)
  Day 182 | 30.31 (17.344)
  Day 266 | 21.69 (11.221)
  Day 350: number analyzed (Participants) | 3
  Day 350 | 39.83 (12.407)
  Day 364: number analyzed (Participants) | 10
  Day 364 | 27.51 (12.901)
  Day 378/392 | 40.65 (15.828)

19. Secondary Outcome: Number of Participants With Positive Anti-drug Antibody (ADA) in Plasma
Description: Baseline was defined as the last non-missing value prior to first dose of study drug (based on date or date/time).
Time Frame: Predose on Days 0 (or Baseline), 56, 98, 140, 182, 266, 350, 364, and at any time on Day 378 or 392
Population: FAS included all participants who received at least 1 dose of IMP. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg q2w or q4w
Number analyzed (Participants) | 12
Participants
  Day 0 (or Baseline) | 0
  Day 56 | 0
  Day 98 | 0
  Day 140: number analyzed (Participants) | 11
  Day 140 | 0
  Day 182 | 0
  Day 266 | 0
  Day 350: number analyzed (Participants) | 3
  Day 350 | 0
  Day 364: number analyzed (Participants) | 10
  Day 364 | 0
  Day 378/392 | 0

20. Secondary Outcome: Number of Participants With TEAEs Related to Clinical Laboratory Tests
Description: A TEAE was defined as any event emerging or manifesting at or after the initiation of treatment with an IP or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the IP or medicinal product. As Pre-specified in the protocol, the treatment emergent adverse events were collected per Period i.e., Treatment Period A, B and Safety follow-up Period. The data is reported as per HAE attack and non-HAE attack per Period. Number of participants with TEAEs related to clinical laboratory tests (hematology, clinical chemistry, coagulation, and urinalysis) were assessed.
Time Frame: From first dose of the study drug up to end of study (EOS) (up to Day 392)
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Period A: Non-HAE: Lanadelumab 300 mg solution, SC, q2w for 26 weeks in Treatment Period A. Non-HAE attack (subset identified in CRF as not reported HAE attack) subset participants were included in this arm.
- Safety Follow-up Period: Non-HAE: Participants who completed the lanadelumab 300 mg regimen in Treatment Period B returned on Day 378 (for participants who chose to roll over into study TAK-743-5007) or Day 392 as follow-up visit for final assessment in the Safety Follow-up Period. Non-HAE attack (subset identified in CRF as not reported HAE attack) subset participants were included in this arm.
Arm/Group | Treatment Period A: Non-HAE | Treatment Period A: HAE | Treatment Period B: Non-HAE | Treatment Period B: HAE | Safety Follow-up Period: Non-HAE | Safety Follow-up Period: HAE
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With TEAEs Related to Vital Signs
Description: A TEAE was defined as any event emerging or manifesting at or after the initiation of treatment with an IP or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the IP or medicinal product. As Pre-specified in the protocol, the treatment emergent adverse events were collected per Period i.e., Treatment Period A, B and Safety follow-up Period. The data is reported as per HAE attack and non-HAE attack per Period. Number of participants with TEAEs related to vital signs (blood pressure (BP), heart rate (HR), body temperature, and respiratory rate) were assessed.
Time Frame: From first dose of the study drug up to end of study (EOS) (up to Day 392)
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period A: Non-HAE | Treatment Period A: HAE | Treatment Period B: Non-HAE | Treatment Period B: HAE | Safety Follow-up Period: Non-HAE | Safety Follow-up Period: HAE
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With TEAEs Related to Electrocardiogram (ECG)
Description: A TEAE was defined as any event emerging or manifesting at or after the initiation of treatment with an IP or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the IP or medicinal product. As Pre-specified in the protocol, the treatment emergent adverse events were collected per Period i.e., Treatment Period A, B and Safety follow-up Period. The data is reported as per HAE attack and non-HAE attack per Period. Number of participants with TEAEs related to 12 lead-ECG were assessed.
Time Frame: From first dose of the study drug up to end of study (EOS) (up to Day 392)
Population: FAS included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period A: Non-HAE | Treatment Period A: HAE | Treatment Period B: Non-HAE | Treatment Period B: HAE | Safety Follow-up Period: Non-HAE | Safety Follow-up Period: HAE
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of the study drug up to end of study (EOS) (up to Day 392)
Description: FAS included all participants who received at least 1 dose of IMP. As Pre-specified in the protocol, the TEAEs were collected per Period i.e., Treatment Period A, B and Safety follow-up Period. The data is reported as per HAE attack and non-HAE attack per Period.
Arm/Group | Treatment Period A: Non-HAE | Treatment Period A: HAE | Treatment Period B: Non-HAE | Treatment Period B: HAE | Safety Follow-up Period: Non-HAE | Safety Follow-up Period: HAE
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/12 | 1/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 10/12 | 7/12 | 9/12 | 8/12 | 0/12 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period A: Non-HAE (N=12) | Treatment Period A: HAE (N=12) | Treatment Period B: Non-HAE (N=12) | Treatment Period B: HAE (N=12) | Safety Follow-up Period: Non-HAE (N=12) | Safety Follow-up Period: HAE (N=12)
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hereditary angioedema (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Treatment Period A: Non-HAE (N=12) | Treatment Period A: HAE (N=12) | Treatment Period B: Non-HAE (N=12) | Treatment Period B: HAE (N=12) | Safety Follow-up Period: Non-HAE (N=12) | Safety Follow-up Period: HAE (N=12)
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 6 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 2 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Infusion site pruritus (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Allergy to chemicals (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Laryngopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Vulvitis (Infections and infestations) | 0/9 | 0/9 | 1/9 | 0/9 | 0/9 | 0/9 — Number of participants at risk in each arm is based on the female population in this study.
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Heat illness (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9 | 0/9 | 1/9 | 0/9 | 0/9 | 0/9 — Number of participants at risk in each arm is based on the female population in this study.
Headache (Nervous system disorders) | 2 | 0 | 2 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0/9 | 0/9 | 1/9 | 0/9 | 0/9 | 0/9 — Number of participants at risk in each arm is based on the female population in this study.
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hereditary angioedema (Congenital, familial and genetic disorders) | 0 | 7 | 0 | 8 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT04180163/Prot_002.pdf
  • Statistical Analysis Plan (2021-01-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT04180163/SAP_003.pdf